CLINICAL TRIAL: NCT00387855
Title: An Outcome Evaluation of the SOS Suicide Prevention Program
Brief Title: An Evaluation of the SOS (Suicide Prevention) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); Patterson Trust (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, ROBERT H. ASELTINE, Professor, Division of Behavioral Sciences and Community Health, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMHS1255; SM 05 014
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Suicide
Keywords: suicide; depression
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): receive SOS program
  Interventions: Behavioral: SOS program

INTERVENTIONS:
Behavioral: SOS program — screening and didactic programming to raise awareness of depression suicidality
  Other Names: Signs of Suicide

SUMMARY:
The purpose of this study was to investigate the impact of the SOS suicide prevention program on help-seeking, attitudes toward depression and suicide, and suicidal behavior among high school students. Current research protocol has extended this evaluation to the Middle School version of SOS.

DETAILED DESCRIPTION:
Three cohorts have participated in outcome evaluations of the SOS suicide prevention program to assess its effects on help-seeking, attitudes toward depression and suicide, and suicidal behavior. The first two cohorts consisted of 25 public state high schools in Massachusetts, Georgia, and Connecticut. The third cohort consisted of 9 middle schools and 10 high schools from outside of Connecticut with high proportions of military dependants.

Hypotheses:

H1: Exposure to the SOS program will be significantly associated with lower rates of suicidal ideation and suicide attempts; greater levels of help-seeking; greater knowledge of and more adaptive attitudes toward depression and suicide; and increased communication with and perceived support from peers.

H2: The reduction in suicide attempts among youths exposed to the program can be explained by increases in knowledge about depression and suicide, more favorable attitudes regarding suicide, and improved communication with and support from peers.

Methods

1. The intervention: The SOS program was presented to students in 2 consecutive classes over a 2 day period, typically in health or social studies classes. The SOS program's teaching materials include a video and a discussion guide. The video includes dramatizations depicting the signs of suicidality and depression, recommended ways to react to someone who is depressed and suicidal, as well as interviews with real people whose lives have been touched by suicide. Students are also asked to complete the Brief Screen for Adolescent Depression (BSAD), a brief screening instrument for depression that is derived from the Diagnostic Interview Schedule for Children IV (Lucas et al., 2001).
2. The sample: The first cohort involved approximately 4000 students in 9 high schools in Columbus Georgia, Hartford Connecticut, and western Massachusetts over a two-year period. The second cohort consisted ove an additional 1100 students were recruited from 16 Technical High Schools in Connecticut. A third cohort consisted of over 600 students from 9 middle schools and 10 high schools from outside of Connecticut with high proportions of military dependants.
3. The research design: The experimental design for the evaluation was a randomized control group design with posttest only data collection. At the beginning of each school year approximately half of the classes of teachers presenting the program were randomly assigned to the treatment group, which received the SOS Prevention Program in the fall/winter of that year; the other half were assigned to the control group, which did not receive the program until the evaluation is completed.

To ascertain the effect of the program on participants' knowledge of and attitudes toward suicide and help seeking behavior, students in both the treatment and control groups were asked to complete a short questionnaire 3 months following implementation of the program. Questionnaires were anonymous. After the outcome evaluation was completed, the group of students who did not receive the program earlier in the school year received the complete SOS Program.

ELIGIBILITY:
Inclusion Criteria:

1. Attendance at school participating in study
2. English speaking youth with parental consent.

Exclusion Criteria:

1.Youth who do not speak and read English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6471 (Actual)
Dates: Start 2001-09; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
suicide attempts | 3 months

SECONDARY OUTCOMES:
knowledge about depression/suicide | 3 months
attitudes about depression/suicide | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Aseltine, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Aseltine RH Jr, DeMartino R. An outcome evaluation of the SOS Suicide Prevention Program. Am J Public Health. 2004 Mar;94(3):446-51. doi: 10.2105/ajph.94.3.446. PMID 14998812
- [Background] Aseltine RH Jr, James A, Schilling EA, Glanovsky J. Evaluating the SOS suicide prevention program: a replication and extension. BMC Public Health. 2007 Jul 18;7:161. doi: 10.1186/1471-2458-7-161. PMID 17640366